CLINICAL TRIAL: NCT06777992
Title: Implementation of Momentum SpineTM: a New 3D Imaging Software for Idiopathic Scoliosis
Status: Not yet recruiting | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Collaborators: Mitacs (Industry); Ministère de l'économie, de l'innovation et de l'énergie du Québec (Unknown); Momentum Health Inc. (Industry); Université de Sherbrooke (Other); Université Clermont-Auvergne, France (Unknown)
Responsible Party: Principal Investigator, Marie Beausejour, Professor-Researcher, St. Justine's Hospital
Other Study IDs: St. Justine's Hospital
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Spine Deformity; Idiopathic Scoliosis
Keywords: Idiopathic scoliosis; Screening; Spine deformity; Progression; Non-invasive 3D scans; Pediatrics
MeSH Terms: conditions — Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control arm: Standard care will be provided to the control arm group. This includes standard 4 to 6-month consultatiosn with the orthopedic surgeons, follow-up standard x-ray (lateral and posterioanterior) examinations, measures of the angle of trunk rotation and Cobb angles, topographic scans performed by the study coordinator using the Momentum Health TM application, at each clincal visits.
- Intervention arm: In addition to the standard care, patients randomized to the Intervention arm of the trial will perform Momentum SpineTM assessment from home at 2-month intervals during the 24-month study follow-up. If a progression is detected using Momentum SpineTM, the participant will be promptly invited to acquire a second set of scans for confirmation. In case of confirmation of the progression using the images from the repeated scans, the scan results will be sent to their local orthopedic surgeon.
  Interventions: Other: Home topographic scans

INTERVENTIONS:
Other: Home topographic scans — Patients randomized to the Intervention arm of the trial will additionally use Momentum SpineTM assessment from home at 2-month intervals. If a progression is detected using Momentum SpineTM the participant will be promptly invited to acquire a second set of scans for confirmation. In case of confirmation of the progression using the images from the repeated scans, the scan results will be sent to their local orthopedic surgeon.
  Groups: Intervention arm

SUMMARY:
Brief Summary

The goal of this clinical trial is to evaluate the implementation of Momentum Spine™, a new 3D imaging software designed to improve the monitoring and management of idiopathic scoliosis in children aged 8-14 years. Idiopathic scoliosis affects 1-3% of the pediatric population and is currently monitored through hospital visits with radiographic imaging every 4-6 months, which exposes patients to cumulative radiation over time. This study explores whether Momentum Spine™ can provide a safer, more accessible alternative by enabling at-home monitoring using clinical photographs taken on smartphones.

The primary questions this study seeks to answer are:

Can Momentum Spine™ accurately predict scoliosis progression, including Cobb angle changes, compared to standard radiographic assessments? Can the use of Momentum Spine™ reduce the number of X-rays required and improve the timing of clinical follow-ups? Does the use of Momentum Spine™ affect patient satisfaction, healthcare utilization, and overall quality of life? This study is a prospective, two-arm randomized controlled trial conducted at CHU Sainte-Justine. Participants will be divided into two groups: the control group will receive standard care, which involves regular clinical visits and radiographic evaluations; the intervention group will use Momentum Spine™ at home, alongside standard care.

Intervention Details

Participants in the intervention group will:

Use the Momentum Spine™ application to capture 3D images of their torso at home every two months. These images will be processed by Momentum Spine™ algorithms to assess curve progression.

Participants will receive notifications and guidance on performing scans at home, supported by the study team to ensure accuracy.

The primary outcomes include clinical measures such as changes in Cobb angle at 1 and 2 years, curve progression of more than 5 degrees, whether the main curve reaches 45 degrees, and the need for surgical referral. Secondary outcomes focus on the accuracy, sensitivity, and specificity of Momentum Spine™, as well as patient-reported measures such as health-related quality of life and satisfaction with care, users' acceptability of the software, healthcare services utilization and pathway costs.

This study also aims to address key challenges in scoliosis care, including reducing radiation exposure, improving follow-up timing to align with growth spurts, and providing equitable access to care for families who may live far from specialty clinics. By validating the performance of Momentum Spine™, this trial has the potential to transform scoliosis management, ensuring safer and more effective care pathways.

DETAILED DESCRIPTION:
This study evaluates the implementation of Momentum Spine™, a novel 3D imaging technology that allows at-home monitoring for patients with idiopathic scoliosis. The objective is to determine whether Momentum Spine™ is as effective as standard radiographic assessments in tracking scoliosis progression while reducing radiation exposure and improving the timing of follow-ups.

Study Rationale & Background:

Idiopathic scoliosis affects approximately 1-3% of the pediatric population and is typically monitored through radiographic imaging every 4-6 months. However, this conventional approach exposes children to significant cumulative radiation over time and is associated with missed opportunities for timely intervention, especially during growth spurts. Momentum Spine™ uses clinical photographs taken on smartphones to generate 3D topographic models of the torso. These models allow for the calculation of the Cobb angle and the detection of curve progression, without requiring frequent radiographs.

Study Design:

This study is a two-arm, randomized controlled trial conducted at CHU Sainte-Justine. Participants will be randomized into two groups:

Control Group: Participants will receive standard care, including radiographic assessments and clinical visits as per current practice.

Intervention Group: Participants will use the Momentum Spine™ 3D imaging software in combination with standard care. They will be asked to perform at-home scans every two months using the Momentum Spine™ application. These scans will be reviewed to track scoliosis progression and compare them to standard clinical evaluations.

Study Objectives:

Primary Objective: Compare the clinical outcomes between participants receiving standard care versus those using Momentum Spine™ in addition to standard care. Key outcomes include changes in Cobb angle and curve progression over a 24-month follow-up.

Secondary Objective: Assess the accuracy of Momentum Spine™'s algorithm compared to radiographic assessments, the proportion of avoidable X-rays, and patient satisfaction during the monitoring period.

Study Procedures:

Participants in the intervention group will receive training on using Momentum Spine™ to capture 3D topographic scans at home every two months. Scans will be submitted through secure servers to Momentum Health for automated analysis. If scans indicate progression of more than 6 degrees in the Cobb angle, participants will be contacted by the research coordinator for confirmation. Results will be shared with the treating orthopedic surgeons to determine whether advanced intervention is required.

The standard of care for both groups will involve clinical visits at regular intervals (every 4-6 months) to assess scoliosis progression and standard clinical management options, including observation, bracing, physiotherapy, or surgical referral when necessary.

Participant Safety:

All participants will follow the standard scoliosis care protocols as recommended by their healthcare providers. Topographic scans and Momentum Spine™ assessments are intended to complement standard care by providing earlier detection of scoliosis progression while minimizing unnecessary radiation exposure. Data privacy and confidentiality are rigorously maintained by encrypting images and anonymizing all scans analyzed by Momentum Health.

Expected Outcomes:

The study will assess whether Momentum Spine™ can accurately predict the Cobb angle of the main curve and be used to detect significant scoliosis progression. It will also explore the number of radiogrpahs that could have been avoided in case of adequate prediction. Additionally, the study will evaluate patient-reported experiences related to satisfaction with care, quality of life, and overall health system use.

This study could lead to a novel, non-invasive approach to scoliosis monitoring and care, with the potential to improve patient outcomes while reducing the risks associated with cumulative radiation exposure from standard imaging methods.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 8 and 14 with a confirmed radiographic diagnosis of Idiopathic Scoliosis who have not undergone spinal nor thoracic surgery.

Exclusion Criteria:

* Patients who may be pregnant. Patients with the existence of a second deformity, or any other neuromuscular condition.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with idiopathic scoliosis diagnosis.
Sampling Method: Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Cobb angle | 1 and 2 years
  The primary outcomes will be clinical progression including: Cobb angle of the main curve at 1 and 2 years of follow up, progression of Cobb angle of more than 5 degrees, whether the main curve reaches 45 degrees during follow-up or whether the patient is referred to surgery.

SECONDARY OUTCOMES:
Performance of the software | All the time
  Secondary outcomes will relate to the performance of the software: accuracy, margin of error, sensitivity, specificity, AUC, overall agreement with radiographs; as well as proportion of accelerated clinical visits and proportion of avoidable x-rays. Additional outcomes will be captured assessing the patient and system related outcomes including: health-related quality of life and satisfaction with care, users' acceptability of the software, healthcare service utilisation and costs of pathways

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Girdler S, Cho B, Mikhail CM, Cheung ZB, Maza N, Kang-Wook Cho S. Emerging Techniques in Diagnostic Imaging for Idiopathic Scoliosis in Children and Adolescents: A Review of the Literature. World Neurosurg. 2020 Apr;136:128-135. doi: 10.1016/j.wneu.2020.01.043. Epub 2020 Jan 16. PMID 31954891
- [Background] Elwyn G, Edwards A, Wensing M, Grol R. Shared Decision Making Measurement using the OPTION instrument. 2005. Accessible from
- [Background] Weinstein SL, Dolan LA, Cheng JC, Danielsson A, Morcuende JA. Adolescent idiopathic scoliosis. Lancet. 2008 May 3;371(9623):1527-37. doi: 10.1016/S0140-6736(08)60658-3. PMID 18456103